CLINICAL TRIAL: NCT02435147
Title: Longitudinal Effects of Denosumab on Trabecular Bone Score and Femur Strength Index
Status: Completed | Type: Observational
Sponsor: HealthEast Care System (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Beth Jorgenson, Clinical Trials Office Program Manager, HealthEast Care System
Other Study IDs: HE 15 03 003
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Osteoporosis; Bone Fracture
MeSH Terms: conditions — Osteoporosis; Fractures, Bone | interventions — Denosumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: denosumab — Patients will receive denosumab 60 mg subcutaneously every six months as part of their standard osteoporosis treatment.
  Other Names: Prolia

SUMMARY:
The purpose of this study is to validate the long-term benefit of denosumab for osteoporosis treatment in a real-world clinical practice setting. We hypothesize that continued therapy (36+months) with denosumab will increase both trabecular bone score (TBS) and femur strength index (FSI) and reduce fracture and other bone health risks among post-menopausal women with osteoporosis.

DETAILED DESCRIPTION:
Bone fractures are a major cause of morbidity and health care expense among patients with osteoporosis.The goal of osteoporosis therapy is to reduce fracture risk. The administration of denosumab 60 mg subcutaneously (SC) every six months has been shown to limit bone turnover, increase bone mineral density (BMD), and reduce the risk for new vertebral, non-vertebral, and hip fractures among postmenopausal women with osteoporosis (Cummings, 2009). Although BMD is an important factor for fracture risk, it does not describe bone microarchitecture, which is related to bone quality and mechanical bone strength. Trabecular bone score (TBS) is an index for bone microarchitecture extracted from anterior-posterior spine dual-energy X-ray absorptiometry (DXA). Previous research has shown TBS to differentiate between women with and without fractures as well as predict future fracture even after adjustment for BMD (Simonelli, Leib, Winzenrieth, & Hans, 2012). In a study of 29,407 Canadian women age 50 years and older at the time of baseline hip and spine DXA, health service records were assessed to determine the incidence of non-traumatic osteoporotic fractures subsequent to BMD testing. Lumbar spine TBS was derived for each DXA examination and blinded to clinical parameters and outcomes. Osteoporotic fractures were identified in 1668 (5.7%) women, including 439 (1.5%) spine and 293 (1.0%) hip fractures. Significantly lower spine TBS and BMD were found in women with major osteoporotic, spine, and hip fractures (p<0.0001). The results of this study suggest that spine TBS is predictive of osteoporotic fractures and provides additional clinical information independent of spine and hip BMD; therefore, combining TBS trabecular texture index with BMD incrementally improves fracture prediction in postmenopausal women (Hans, Goertzen, Krieg, & Leslie, 2011).

Clinical research has demonstrated the positive effect of denosumab on TBS over time. In a randomized, double-blind, placebo-controlled trial of 215 postmenopausal women with low BMD at the spine or total hip, denosumab (60mg SC every 6 months) was found to increase lumbar spine QCT, DXA, and TBS at 12 months compared to placebo or alendronate (Thomas, 2013). In another study conducted by McClung et al, postmenopausal women with osteoporosis who received denosumab were found to have significant increases in TBS, independent of BMD, at 36 months compared to baseline and placebo (McClung, Lippuner, Brandi, Kaufman, Zanchetta, & Krieg, 2012).

Femur strength index (FSI), which is a measure of femoral bone density, structure, and strength, has also been shown to predict hip fracture independent of bone density and hip axis length. In a study which compared FSI in a group of women age 50 years and older with and without hip fracture (365 with prior hip fracture and 2,141 controls), FSI was found to be significantly lower in the fracture group, after adjusting for T score and hip axis length (Faulkner, et al., 2006). Like TBS, FSI can be obtained from femur DXA measurements using modern software.

This is a single-site, open-label, non-randomized, observational study designed to assess the change in TBS and FSI at 36 months. among post-menopausal women with osteoporosis taking denosumab. All patients included in this study are under the medical care of the principal investigator. Subjects will enter the study once they have completed 36 months of treatment with denosumab and have evaluable DXA scans. Medical records will be retrospectively reviewed and percent change in TBS and FSI scores will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following inclusion criteria to be eligible for study entry:

  * Post-menopausal female with diagnosed osteoporosis
  * Age 40-90 years
  * Completed 36 months of denosumab therapy (SQ; 60mg every 6 months) but not yet received the 42 month injection
  * Availability of DXA scans at the study-required time points, including the willingness of subjects to undergo a DXA evaluation at 36 months, if required
  * Provided written informed consent

Exclusion Criteria:

* Patients will be excluded from this study for any of the following reasons:

  * Received denosumab injections for less than 36 months
  * Patients who have missed more than 1 dose of denosumab in a 36 month period
  * Contra-indicated for treatment with denosumab
  * History of rheumatoid arthritis
  * Current diagnosis of hyperparathyroidism; hyperthyroidism; osteomalacia, or other known diseases that can affect bone
  * In the opinion of the investigator, have any kind of disorder that may compromise the ability of the subject to provide written informed consent

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll postmenopausal women between the ages of 40 and 90 years who have completed a minimum of 36 months of denosumab therapy for the treatment of osteoporosis.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Simonelli, MD, Principal Investigator — HealthEast Care System
Locations (1):
- HealthEast Care System, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a single-site, non-randomized observational study of post-menopusal women between the ages of 40 and 90 years who completed a minimum of 36 months of denosumab therapy for the treatment of osteoporosis and had evaluable DXA scans. Women were recruited to participate from a single clinical practice site between March 2015 and March 2016.
Groups:
- Denosumab: This is a single-site, open-label, non-randomized observational study of postmenopausal women with osteoporosis being actively treated with denosumab. All participants received denosumab as part of their standard of care osteoporosis therapy.
Period: Overall Study
Arm/Group | Denosumab
Started | 86
Completed | 75
Not Completed | 11
Not completed — non-evaluable DXA scan | 11

BASELINE CHARACTERISTICS:
Arm/Group | Denosumab
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 75
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 75
Trabecular Bone Score [Mean (Standard Deviation); unit: units on a scale] — Trabecular Bone Score (TBS) is an index for bone micro-architecture extracted from anterior-posterior spine dual-energy X-ray absorptiometry (DXA) images. TBS quantifies local variations in pixel intensities and is derived from the experimental variogram obtained from the gray levels of a DXA image. As noted in the Journal of Bone Mineral Research Volume 29, Issue 3, March 2014, pages 518-530, "TBS> or = 1.350 is considered to be normal; TBS between 1.200 and 1.350 is considered to be consistent with partially degraded microarchitecture, and TBS </=1.200 defines degraded microarchitecture".
  units on a scale | 1.257 (0.09)
Femur Strength Index [Mean (Standard Deviation); unit: units on a scale] — Femur strength index (FSI) is a measure of femoral bone density, structure and strength obtained from DXA measurements using modern software. FSI provides an index for hip strength by combining bone mineral density, femur geometry, age, height, and weight.This index is not anchored in definite values, but rather is derived from the following equation: Hip Strength Index= strength/stress where, strength=185-0.34 (age-45); Age>45 years. Stress=moment*y/CSM I+ force/CSA. Higher values indicate greater hip strength.
  units on a scale | 1.291 (0.287)
Lumbar Spine Bone Mineral Density [Mean (Standard Deviation); unit: g/cm^2] — Lumbar bone mineral density is measured in g/cm^2 and is dependent on such factors such as an individual's age, height, weight and ethnicity.
  g/cm^2 | 0.931 (0.132)
Femoral Neck Bone Mineral Density [Mean (Standard Deviation); unit: g/cm^2] — Femoral neck bone mineral density is measured in g/cm^2 and is dependent on such factors as an individual's age, height, weight and ethnicity.
  g/cm^2 | 0.717 (0.070)
Total Femur Bone Mineral Density [Mean (Standard Deviation); unit: g/cm^2] — Total femur bone mineral density is measured in g/cm^2 and is dependent on factors such as an individual's age, height, weight, and ethnicity.
  g/cm^2 | 0.746 (0.079)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Change in Mean Trabecular Bone Score
Description: Proportion of change in mean trabecular bone score at 36 months following denosumab initiation
Time Frame: Baseline and 36 months
Measure: Mean (Standard Deviation); unit: Proportion of change
Arm/Group | Denosumab
Number analyzed (Participants) | 75
Proportion of change | .00238 (0.0422)

2. Secondary Outcome: Proportion of Change in Mean Femur Strength Index Score
Description: Proportion of change in mean Femur Strength Index Score at 36 months following denosumab initiation
Time Frame: Baseline and 36 months
Measure: Mean (Standard Deviation); unit: Proportion of change
Arm/Group | Denosumab
Number analyzed (Participants) | 75
Proportion of change | .0838 (.2208)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Denosumab
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

LIMITATIONS AND CAVEATS:
This is a small observational study of Caucasian women in a single, Midwest clinical practice. The results cannot be generalized to the broader population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No